CLINICAL TRIAL: NCT05760846
Title: Exploring the Neural Substrates of Proximal and Distal Bimanual Motor Skill Learning Through Robotics and Multimodal Brain Imaging
Brief Title: Bimanual Motor Skill Learning in Acute Stroke
Acronym: MLAS4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Principal Investigator, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Bim-MSkL acute
Record Dates: First submitted 2023-02-22; First posted 2023-03-08 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Acute; Stroke, Subacute
Keywords: Motor Skill Learning; Upper limb; Acute stroke; Rehabilitation; Subacute stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Not aware being of the different versions of the tasks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimanual Circuit version 1 (Experimental): Training on the REAplan® robot with a serious game based on proximal motor skill learning (bim-MSkL) with the bimanual version 1 of the Circuit task and training on the Dextrain Manipulandum with a serious game based on distal bim-MSkL
  Interventions: Device: REAplan®; Device: Dextrain Manipulandum®
- Bimanual Circuit version 2 (Experimental): Training on the REAplan® robot with a serious game based on motor skill learning (MSkL) with bimanual version 2 of the Circuit task and training on the Dextrain Manipulandum with a serious game based on distal bim-MSkL
  Interventions: Device: REAplan®; Device: Dextrain Manipulandum®

INTERVENTIONS:
Device: REAplan® — motor skill learning with the REAplan® rehabilitation robot, to be performed with both arms
Device: Dextrain Manipulandum® — motor skill learning with the Dextrain Manipulandum® dexterity tool to be performed with both hands

SUMMARY:
The subacute phase of stroke provides a window into how a lesion perturbs sensorimotor functions prior to reorganisation driven by plasticity and neurorehabilitation. The recovery from motor impairment has been extensively studied, but it is currently unknown whether motor skill learning (MSkL) is enhanced or impaired during acute stroke, especially bimanual motor skill learning (bim-MSkL), which likely requires more motor-attentional-cognitive resources than unimanual MSkL.

The goals of this project are: to determine the neural substrates critical to achieve proximal and distal bimanual motor skill learning (bim-MSkL) by specifying whether (sub)acute stroke to different brain areas (cortical and subcortical) induce specific deficits in bimanual and/or distal bim-MSkL, which behavioral components are involved in bim-MSkL, and whether damage to the motor, sensory and inter-hemispheric pathways specifically impairs proximal and/or distal bim-MSkL.

DETAILED DESCRIPTION:
Over 3 consecutive days, the patients will be evaluated and will train on the rehabilitation robot REAplan® (http://www.axinesis.com/) to assess proximal bim-MSkL and on the manual dexterity tool Dextrain Manipulandum (https://www.dextrain.com/) to assess distal bim-MSkL.

For proximal bim-MSkL, patients will train over the 3 days on the serious game Circuit on the bimanual REAplan® and will be randomised to two different bimanual versions. By this means, the investigators will explore the components of bim-MSkL in acute stroke patients.

The motor skill learning setup (Circuit) that was developed and successfully used in healthy individuals and stroke patients has already been implemented in the REAplan® environment and will be used as innovative serious games based on a speed/accuracy trade-off (SAT), allowing a detailed analysis of motor skill learning components (speed, accuracy, SAT, movement smoothness, dynamics...). For the serious game Circuit, who based on motor skill learning, the subjects will have to practice a complex circuit and move a cursor as quickly and accurately as possible by controlling the handles of the robot with both arms.

For distal bim-MSkL, patients will train on a complex sequence of finger movements involving both hands. Each day, several successive repetitions of the sequence will be displayed, corresponding to one block. 3 to 6 blocks will be repeated, each separated by 30 sec of rest. After training on the third day, a new sequence will be repeated for 3 blocks to assess generalization.

To explore the role of different brain structures in bim-MskL, Voxel-based Lesion Symptom Mapping (VLSM) based on high-resolution brain magnetic resonance imaging (MRI) scans, will be used to analyse the relationship between tissue damage and proximal/distal bim-MskL scores on a voxel-by-voxel basis.

Diffusion Tensor Imaging (DTI) will quantify the integrity of several white matter tracts, allowing through correlation analyses to unveil the white matter tracts crucial to achieve proximal and/or distal bim-MskL.

In addition, several "classical" clinical scales and tests will be used to evaluate overall motor-sensory-cognitive functions.

In addition to the (sub)acute stroke patients, a group of healthy individuals who will not undergo MRI (n=60) will be enrolled as control group. Subjects in this group will also be randomized 1/1 in the two versions of the bimanual Circuit task on the REAplan® robot.

ELIGIBILITY:
ACUTE STROKE PATIENTS:

Inclusion Criteria:

* acute stroke (< 21 days)
* aged 18-90 years
* with a demonstrated stroke (ischemic or hemorrhagic) lesion on brain imaging

Exclusion Criteria:

* " classical " contre-indication to MRI (non-MR-compatible pacemaker, pregnancy, non-MR-compatible implanted devices, claustrophobia, etc ...)
* difficulty in understanding or executing commands
* drug/alcohol abuse
* severe aphasia / cognitive deficits interfering with study
* inability to complete the tasks (i.e. full paralysis of the arm)
* multiple strokes / dementia / psychiatric condition

HEALTHY INDIVIDUALS:

Inclusion Criteria:

• 18-90 years

Exclusion Criteria:

* medical history with a previous stroke / relevant neurological deficit
* drug/alcohol abuse
* psychiatric condition/ dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
bimanual Speed/Accuracy Trade-off (bi-SAT), bimanual Speed/Accuracy Trade-off measured by the REAplan® robot | change between baseline (Day 1) and after training (Day 3)
  bimanual Speed/Accuracy Trade-off: mathematical computation of the relationship between speed and accuracy
bimanual Coordination factor (bi-CO), bimanual Coordination factor measured by the REAplan® robot | change between baseline (Day 1) and after training (Day 3)
  bimanual Coordination factor, mathematical measure of the phase coherence between speeds of both arms
bi-Force, bimanual force measured by the REAplan® robot | change between baseline (Day 1) and after training (Day 3)
  bimanual forces, forces exerted in the wrong direction by each arm (Newtons)
Root Mean Square Error (RMSE), bimanual root mean square error measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  Tracking error between the actual applied force and the target force
Bimanual Dexterity Coordination Index measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  bimanual Coordination factor, mathematical measure of the phase coherence between speeds of both thumb-index clamps

SECONDARY OUTCOMES:
Reaction time measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  time between the target appearance and when the force applied exceeds threshold
Rise time measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  time between the reaction time and reaching the plateau
Coactivation measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  binary measure of unasked fingers activated above the force threshold
Hold time measured by the Dextrain Manipulandum | change between baseline (Day 1) and after training (Day 3)
  time of plateau maintenance
Voxel-based Lesion Symptom Mapping (VLSM) | Baseline
  Diffusion Weighted Imaging (DWI)
Diffusion Tensor Imaging (DTI) | Baseline
  Fractional Anisotropy
Fugl Meyer Upper Extremity Test (FMA-UE) | Day1
  Tests impairments of the upper limb after stroke. Range: 0-66. A higher score means less impairment.
Arm Motor Ability (AMA) test | Day 1
  Measure disabilities of the upper limb after stroke. Range: 0-100. A higher score means less disabilities in activities of daily living.
Montreal Cognitive Assessment (MoCA) | Day 1
  Tests the short-term memory, visuospatial skills, executive functions, attention, concentration, working memory, language and orientation in time and space. Range: 0-30, higher score means no cognitive impairment.
Fatigue Visual Analog Scale (VAS) | Day 1
  Visual Analog Scale to evaluate fatigue = a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Range : 0- 10. A higher score means a higher level of fatigue.
Shoulder Abduction Finger Extension (SAFE) test | Day 1
  A prognostic determinant of the function of the hemiparetic upper limb (UL) after a stroke. For each of the 2 subitems, the range is 0-5. A score of 5 means normal power. A score of 0 means no contraction possible.
Modified Ashworth Scale (mAS) | Day 1
  clinical measure of spasticity. For each of the 8 subitems, the range is 0-4. A higher score means a higher level of spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vandermeeren, MD, PhD, Principal Investigator — UCLouvain IONS
Locations (2):
- Belgium (2):
  - CHU UCL Namur, Yvoir, Namur
  - University Hospital CHU Dinant Godinne UCL, Yvoir

IPD SHARING:
Plan to Share IPD: Yes
Data Management Plan REDCap
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during the beginning of the study and for 20 years.
Access Criteria: Login user of the Hospital of CHU UCL Namur -Site Godinne